CLINICAL TRIAL: NCT07028593
Title: Effects of Ciprofol on Myocardial Injury After Non-cardiac Surgery (CP-MINS) in Patients Undergoing Video-Assisted Thoracoscopic Surgery: A Randomized, Double-Blind, Propofol-Controlled, Multicenter Trial
Brief Title: Effects of Ciprofol on Myocardial Injury After Non-cardiac Surgery in Video-Assisted Thoracoscopic Surgery
Acronym: CP-MINS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Ailin Luo, Department of Anesthesiology, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TJ-IRB202502133
Record Dates: First submitted 2025-05-29; First posted 2025-06-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Injury; Thoracic Diseases; Thoracoscopic Surgery
Keywords: Myocardial Injury after non-cardiac surgery; Ciprofol; propofol; Video-Assisted Thoracoscopic Surgery; lung tumor
MeSH Terms: conditions — Thoracic Diseases; Lung Neoplasms | interventions — Propofol; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; HSK3486

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study blinded the efficacy assessors (rather than the anesthesiologists administering the anesthesia) and the participants, with the double-blind status maintained throughout the study period.
  1. Blinding of efficacy assessors: In this study, a designated study coordinator was responsible for maintaining and distributing randomization numbers, preparing study drugs, and coordinating information among anesthesiologists. Anesthesiologists completed preoperative visits and collected preoperative patient data; efficacy evaluators were only responsible for patient follow-up and data entry of postoperative test results, without participating in the process of anesthesia administration or management. Anesthesiologists administered drugs based on patients' body weights.
  2. Blinding of participants: participants were unaware of their group assignments and medication administration during the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ciprofol group (Experimental): Slowly administer sufentanil 0.2 μg/kg to 0.7 μg/kg via intravenous injection; cis-atracurium 0.15 mg/kg to 0.20 mg/kg; Ciprofol 0.4 ml/kg to 0.6 ml/kg via slow intravenous injection. The injection time for all drugs is 2 minutes.
  Interventions: Drug: ciprofol
- propofol group (Active Comparator): Slowly administer sufentanil 0.2 μg/kg to 0.7 μg/kg via intravenous injection; cis-atracurium 0.15 mg/kg to 0.20 mg/kg; propofol injection 0.1 ml/kg to 0.25 ml/kg slowly via intravenous injection. The injection time for all drugs is 2 minutes.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Using as sedative agents in the total intravenous anesthesia in video-assisted thoracoscopic aurgery in propofol group.
  Arms: propofol group
Drug: ciprofol — Using as sedative agents in the total intravenous anesthesia in video-assisted thoracoscopic aurgery in ciprofol group.
  Other Names: HSK3486
  Arms: ciprofol group

SUMMARY:
Myocardial injury after noncardiac surgery (MINS) refers to postoperative elevation of cardiac troponin (cTn) levels caused by underlying ischemic mechanisms (i.e., coronary artery supply-demand imbalance or atherosclerotic thrombosis) without obvious non-ischemic causes (such as pulmonary embolism), with at least one cTn concentration exceeding the 99th percentile of the test reference upper limit, regardless of whether clinical symptoms and ECG changes are present. MINS, including myocardial infarction and ischemic myocardial injury, typically occurs within 30 days after surgery, most commonly within the first 2 postoperative days. It is an independent risk factor for 30-day postoperative mortality and is also closely associated with increased risk of mortality and vascular complications within 2 years . MINS is a common cardiovascular complication after thoracic surgery. Therefore, reducing the incidence of MINS in non-cardiac thoracic surgery to improve patient outcomes is a critical issue in anesthetic management for thoracic surgery.

Ciprofol is a Class 1 innovative drug independently developed in China with global intellectual property rights. Currently, Ciprofol has completed Phase III clinical trials in China and the United States; its approved indications in China include sedation or anesthesia for various diagnostic procedures, general anesthesia for surgical operations, and sedation during intensive care unit (ICU) stays. Completed drug clinical trials and published clinical trial data of Ciprofol indicate that it can better maintain circulatory stability and ideal anesthetic depth during anesthesia induction and maintenance, making it a promising intravenous general anesthetic alternative to propofol.

Maintaining hemodynamic stability is an important measure to reduce cardiovascular complications during the perioperative period. Given the good circulatory stability and sedative efficacy of Ciprofol, this study aims to investigate the impact of Ciprofol on MINS in non-cardiac thoracic surgery.

DETAILED DESCRIPTION:
Lung cancer ranks first in both incidence and mortality among malignant tumors in China. In 2022, there were 1,060,600 new lung cancer cases, accounting for 22.0% of all malignant tumors, and 733,300 deaths, accounting for 28.5% of all malignant tumor deaths. Radical surgical resection is the recommended preferred treatment for stage I and II non-small cell lung cancer. Video-assisted thoracoscopic surgery (VATS) for anatomic lung resection has better safety and long-term efficacy than traditional surgical methods, with more than 73.7% of lung cancer surgeries in China using thoracoscopic approaches. Thoracic surgery easily induces significant perioperative hemodynamic fluctuations, increasing the risk of perioperative cardiovascular and cerebrovascular complications, thus posing great challenges to perioperative anesthetic safety and long-term patient outcomes.

Myocardial injury after noncardiac surgery (MINS) refers to postoperative elevation of cardiac troponin (cTn) levels caused by underlying ischemic mechanisms (i.e., coronary artery supply-demand imbalance or atherosclerotic thrombosis) without obvious non-ischemic causes (such as pulmonary embolism), with at least one cTn concentration exceeding the 99th percentile of the test reference upper limit, regardless of whether clinical symptoms and ECG changes are present. MINS, including myocardial infarction and ischemic myocardial injury, typically occurs within 30 days after surgery, most commonly within the first 2 postoperative days. It is an independent risk factor for 30-day postoperative mortality and is also closely associated with increased risk of mortality and vascular complications within 2 years. MINS is a common cardiovascular complication after thoracic surgery; the COP-AF study found that the incidence of MINS in non-cardiac thoracic surgery is 20.3% . Therefore, reducing the incidence of MINS in non-cardiac thoracic surgery to improve patient outcomes is a critical issue in anesthetic management for thoracic surgery.

Severe hemodynamic fluctuations are one of the important causes of perioperative induction of MINS, thus maintaining hemodynamic stability is a critical step to reduce MINS. Propofol is the most commonly used drug for anesthesia induction and maintenance in clinical practice, with advantages such as rapid onset, strong sedative efficacy, and quick recovery. However, due to its significant circulatory inhibitory effects, the incidence of intraoperative hypotension induced and maintained by propofol in patients without cardiovascular diseases is 25%-40%, increasing the risk of perioperative hypotension and adverse cardiovascular events, which poses great challenges to anesthetic management. Additionally, 80% of patients receiving propofol experience injection pain of varying degrees, which also reduces patient comfort during treatment. Therefore, developing a sedative with both good sedative efficacy and no or low circulatory inhibition has long been a desirable goal for anesthesiologists.

Ciprofol is a Class 1 innovative drug independently developed in China with global intellectual property rights. Its molecular structure is an analog of propofol (2,6-diisopropylphenol). Both Ciprofol and propofol act on γ-aminobutyric acid type A (GABA-A) receptors, causing hyperpolarization of GABAergic neurons, reducing the success rate of action potential generation, and achieving inhibition of the central nervous system to produce short and rapid sedative or anesthetic effects. Pharmacologically, Ciprofol not only retains the characteristics of propofol such as rapid onset, rapid elimination, and high sedative efficacy but also has a higher drug cost-effectiveness ratio and therapeutic index (in mouse experiments, the median effective dose for sedation of Ciprofol is 1.5 mg/kg, the median lethal dose is 9.9 mg/kg, and the therapeutic index is 6.6, while that of propofol is only 2.8). Furthermore, due to the lower drug concentration in the aqueous phase of the Ciprofol emulsion, the risk of injection pain is much lower than that of propofol, improving treatment comfort. Currently, Ciprofol has completed Phase III clinical trials in China and the United States; its approved indications in China include sedation or anesthesia for various diagnostic procedures, general anesthesia for surgical operations, and sedation during intensive care unit (ICU) stays. Completed drug clinical trials and published post-marketing clinical trial data of Ciprofol indicate that it can better maintain circulatory stability and ideal anesthetic depth during anesthesia induction and maintenance, making it a promising intravenous general anesthetic alternative to propofol.

Maintaining hemodynamic stability is an important measure to reduce cardiovascular complications during the perioperative period. Given the good circulatory stability and sedative efficacy of Ciprofol, this study aims to investigate the impact of Ciprofol on MINS in non-cardiac thoracic surgery.

After data collection, full Analysis Set (FAS): A population derived by minimally and reasonably excluding certain cases under the principle of Intention-to-Treat (ITT), where cases included in the FAS should not seriously violate the inclusion criteria. FAS will be used for the analysis of baseline data and primary efficacy endpoints.

Per-Protocol Set (PPS): All cases that comply with the trial protocol, are well-tolerated (patients who completed PED procedures), and have completed the content specified in the case report form. PPS is used for the analysis of primary efficacy endpoints.

Safety Set (SS): Refers to the actual data of subjects who received at least one dose of treatment after randomization and have recorded safety indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for elective video-assisted thoracoscopic (VATS)-assisted thoracic surgery (lobectomy, segmentectomy, wedge resection of two or more lung tissues, mediastinal tumor resection) under general anesthesia;
2. Aged 45 to 80 years (inclusive) at the time of randomization;
3. Expected postoperative hospital stay of ≥3 days;
4. Signed a written informed consent to participate in the study.

Exclusion Criteria:

1. Patients allergic to propofol, Ciprofol, or analogs of drug excipient components (soybeans, eggs, milk);
2. Patients with unstable angina;
3. Patients with congestive heart failure or hemodynamic instability requiring vasopressor agents;
4. Patients with severe COPD (FEV1 < 1 L);
5. Glomerular filtration rate [eGFR] < 30 mL/min/1.73m²;
6. Patients with severe hepatic dysfunction (ALT or AST elevation exceeding 1.5 times the upper limit of normal);
7. Male or female patients planning to conceive within the next 3 months;
8. Pregnant or lactating female patients;

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1058 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of myocardial Injury after non-cardiac surgery | Within the first 30 days after surgery
  Myocardial injury after noncardiac surgery is defined by elevated postoperative cardiac troponin concentrations that exceed the 99th percentile of the upper reference limit of the assay and are attributable to a presumed ischemic mechanism, with or without concomitant symptoms or signs

SECONDARY OUTCOMES:
The proportion of new-onset atrial fibrillation | within hospitalized stay after anesthesia induction
  diagnosed by 12 lead ECG.
The proportion of new-onset atrial fibrillation | perioperatively
  diagnosed by 12 lead ECG.
The proportion of new-onset non-atrial fibrillation arrhythmia | perioperatively
  diagnosed by 12 lead ECG.
The incidence and duration of perioperative hypotension | between anesthesia induction and postoperative first 24 hour
  assessing the effect of interventions on cardiovascular stability
30-day postoperative mortality rate | Within the first 30 days after surgery
  assessing the survival outcome
New-onset myocardial infarction | Within the first 30 days after surgery
  assessing the cardiovascular complications

OTHER OUTCOMES:
pain on injection of drugs | During anesthesisa induction
  NRS was used to evaluate the pain intensity
the duration of bis>60 or bis <40 | intraoperatively
  assessing the sedative effcacy and avoding intraoperative awareness
Spontaneous respiration recovery time | intraoperatively
  assessing the effect of interventions rescovery time
ermergence time | intraoperatively
  assessing the effect of interventions rescovery time
Intraoperative dosage of vasoactive drug | from anesthesia induction to PACU
  text the species and dosage of drugs
postoperative delirium | during stay in PACU
  assess with CAM-ICU
The time stay in PACU | during stay in PACU
  assessing the effect of interventions rescovery quality
the incidence of postoperative nausen and vomitting | perioperatively
  assessing the effect of interventions on PONV
QoR-15 | postoperatively day 1 and day3
  using Chinsese edition QoR-15
Brice screening | one time in PACU and anther one with postoperative day 1
  To assess intraoperative awareness
time to MOAA/S 0 | from the injection of propofol or ciprofol
  Assessing induction time duration

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Wuhan, China

REFERENCES:
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Circulation. 2018 Nov 13;138(20):e618-e651. doi: 10.1161/CIR.0000000000000617. No abstract available. PMID 30571511
- [Background] Lopez J, Borzak S. In noncardiac thoracic surgery, low-dose colchicine did not reduce AF or myocardial injury after noncardiac surgery at 14 d. Ann Intern Med. 2024 Jan;177(1):JC3. doi: 10.7326/J23-0103. Epub 2024 Jan 2. PMID 38163371
- [Background] Conen D, Ke Wang M, Popova E, Chan MTV, Landoni G, Cata JP, Reimer C, McLean SR, Srinathan SK, Reyes JCT, Grande AM, Tallada AG, Sessler DI, Fleischmann E, Kabon B, Voltolini L, Cruz P, Maziak DE, Gutierrez-Soriano L, McIntyre WF, Tandon V, Martinez-Tellez E, Guerra-Londono JJ, DuMerton D, Wong RHL, McGuire AL, Kidane B, Roux DP, Shargall Y, Wells JR, Ofori SN, Vincent J, Xu L, Li Z, Eikelboom JW, Jolly SS, Healey JS, Devereaux PJ; COP-AF Investigators. Effect of colchicine on perioperative atrial fibrillation and myocardial injury after non-cardiac surgery in patients undergoing major thoracic surgery (COP-AF): an international randomised trial. Lancet. 2023 Nov 4;402(10413):1627-1635. doi: 10.1016/S0140-6736(23)01689-6. Epub 2023 Aug 25. PMID 37640035
- [Background] Zucker M, Kagan G, Adi N, Ronel I, Matot I, Zac L, Goren O. Changes in mean systemic filling pressure as an estimate of hemodynamic response to anesthesia induction using propofol. BMC Anesthesiol. 2022 Jul 22;22(1):234. doi: 10.1186/s12871-022-01773-8. PMID 35869445
- [Background] de Wit F, van Vliet AL, de Wilde RB, Jansen JR, Vuyk J, Aarts LP, de Jonge E, Veelo DP, Geerts BF. The effect of propofol on haemodynamics: cardiac output, venous return, mean systemic filling pressure, and vascular resistances. Br J Anaesth. 2016 Jun;116(6):784-9. doi: 10.1093/bja/aew126. PMID 27199311
- [Background] Jalota L, Kalira V, George E, Shi YY, Hornuss C, Radke O, Pace NL, Apfel CC; Perioperative Clinical Research Core. Prevention of pain on injection of propofol: systematic review and meta-analysis. BMJ. 2011 Mar 15;342:d1110. doi: 10.1136/bmj.d1110. PMID 21406529
- [Background] Gan TJ, Bertoch T, Habib AS, Yan P, Zhou R, Lai YL, Liu X, Essandoh M, Daley WL, Gelb AW. Comparison of the Efficacy of HSK3486 and Propofol for Induction of General Anesthesia in Adults: A Multicenter, Randomized, Double-blind, Controlled, Phase 3 Noninferiority Trial. Anesthesiology. 2024 Apr 1;140(4):690-700. doi: 10.1097/ALN.0000000000004886. PMID 38150544
- [Background] Qin L, Ren L, Wan S, Liu G, Luo X, Liu Z, Li F, Yu Y, Liu J, Wei Y. Design, Synthesis, and Evaluation of Novel 2,6-Disubstituted Phenol Derivatives as General Anesthetics. J Med Chem. 2017 May 11;60(9):3606-3617. doi: 10.1021/acs.jmedchem.7b00254. Epub 2017 Apr 28. PMID 28430430
- [Background] Liang P, Dai M, Wang X, Wang D, Yang M, Lin X, Zou X, Jiang K, Li Y, Wang L, Shangguan W, Ren J, He H. Efficacy and safety of ciprofol vs. propofol for the induction and maintenance of general anaesthesia: A multicentre, single-blind, randomised, parallel-group, phase 3 clinical trial. Eur J Anaesthesiol. 2023 Jun 1;40(6):399-406. doi: 10.1097/EJA.0000000000001799. Epub 2023 Jan 19. PMID 36647565
- [Background] Wang X, Wang X, Liu J, Zuo YX, Zhu QM, Wei XC, Zou XH, Luo AL, Zhang FX, Li YL, Zheng H, Li H, Wang S, Wang DX, Guo QL, Liu CM, Wang YT, Zhu ZQ, Wang GY, Ai YQ, Xu MJ. Effects of ciprofol for the induction of general anesthesia in patients scheduled for elective surgery compared to propofol: a phase 3, multicenter, randomized, double-blind, comparative study. Eur Rev Med Pharmacol Sci. 2022 Mar;26(5):1607-1617. doi: 10.26355/eurrev_202203_28228. PMID 35302207
- [Background] Zeng Y, Wang DX, Lin ZM, Liu J, Wei XC, Deng J, Liu YF, Ma EL, Yang MC, Zheng H, Yu XD, Guo QL, Guan YJ. Efficacy and safety of HSK3486 for the induction and maintenance of general anesthesia in elective surgical patients: a multicenter, randomized, open-label, propofol-controlled phase 2 clinical trial. Eur Rev Med Pharmacol Sci. 2022 Feb;26(4):1114-1124. doi: 10.26355/eurrev_202202_28101. PMID 35253166
- [Background] Liu Y, Yu X, Zhu D, Zeng J, Lin Q, Zang B, Chen C, Liu N, Liu X, Gao W, Guan X. Safety and efficacy of ciprofol vs. propofol for sedation in intensive care unit patients with mechanical ventilation: a multi-center, open label, randomized, phase 2 trial. Chin Med J (Engl). 2022 May 5;135(9):1043-1051. doi: 10.1097/CM9.0000000000001912. PMID 34924506
- [Background] Luo Z, Tu H, Zhang X, Wang X, Ouyang W, Wei X, Zou X, Zhu Z, Li Y, Shangguan W, Wu H, Wang Y, Guo Q. Efficacy and Safety of HSK3486 for Anesthesia/Sedation in Patients Undergoing Fiberoptic Bronchoscopy: A Multicenter, Double-Blind, Propofol-Controlled, Randomized, Phase 3 Study. CNS Drugs. 2022 Mar;36(3):301-313. doi: 10.1007/s40263-021-00890-1. Epub 2022 Feb 14. PMID 35157236
- [Background] Li J, Wang X, Liu J, Wang X, Li X, Wang Y, Ouyang W, Li J, Yao S, Zhu Z, Guo Q, Yu Y, Meng J, Zuo Y. Comparison of ciprofol (HSK3486) versus propofol for the induction of deep sedation during gastroscopy and colonoscopy procedures: A multi-centre, non-inferiority, randomized, controlled phase 3 clinical trial. Basic Clin Pharmacol Toxicol. 2022 Aug;131(2):138-148. doi: 10.1111/bcpt.13761. Epub 2022 Jun 10. PMID 35653554
- [Background] Teng Y, Ou M, Wang X, Zhang W, Liu X, Liang Y, Li K, Wang Y, Ouyang W, Weng H, Li J, Yao S, Meng J, Shangguan W, Zuo Y, Zhu T, Liu B, Liu J. Efficacy and safety of ciprofol for the sedation/anesthesia in patients undergoing colonoscopy: Phase IIa and IIb multi-center clinical trials. Eur J Pharm Sci. 2021 Sep 1;164:105904. doi: 10.1016/j.ejps.2021.105904. Epub 2021 Jun 8. PMID 34116176
- [Result] Puelacher C, Lurati Buse G, Seeberger D, Sazgary L, Marbot S, Lampart A, Espinola J, Kindler C, Hammerer A, Seeberger E, Strebel I, Wildi K, Twerenbold R, du Fay de Lavallaz J, Steiner L, Gurke L, Breidthardt T, Rentsch K, Buser A, Gualandro DM, Osswald S, Mueller C; BASEL-PMI Investigators. Perioperative Myocardial Injury After Noncardiac Surgery: Incidence, Mortality, and Characterization. Circulation. 2018 Mar 20;137(12):1221-1232. doi: 10.1161/CIRCULATIONAHA.117.030114. Epub 2017 Dec 4. PMID 29203498
- [Result] Ruetzler K, Smilowitz NR, Berger JS, Devereaux PJ, Maron BA, Newby LK, de Jesus Perez V, Sessler DI, Wijeysundera DN. Diagnosis and Management of Patients With Myocardial Injury After Noncardiac Surgery: A Scientific Statement From the American Heart Association. Circulation. 2021 Nov 9;144(19):e287-e305. doi: 10.1161/CIR.0000000000001024. Epub 2021 Oct 4. PMID 34601955